CLINICAL TRIAL: NCT06530992
Title: The Effect of Tucking on Semen Quality of Adult Trans Women Compared to Semen Quality of Trans Women Who do Not Tuck - a Case Control Study
Brief Title: The Effect of Tucking on Semen Quality of Adult Trans Women
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1162/2024V2.0
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Transgender; Gender Incongruence; Fertility Issues
MeSH Terms: conditions — Gender Dysphoria; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- tucking: trans women who practice tucking
  Interventions: Other: tucking break
- no tucking: trans women who do not practice tucking

INTERVENTIONS:
Other: tucking break — All participants will provide a semen sample for sperm analysis after 2-7 days of abstinence from ejaculation, a venous blood sample will be taken at the same time, and quality of life will be assessed using a questionnaire.
  Participants in the study group are then asked to refrain from tucking or wearing tight underwear for at least 73 days. At least 73 days (10.5 weeks) after the first spermiogram, another semen collection is scheduled after 2-7 days of abstinence from ejaculation for the preparation of a spermiogram, a venous blood sample is taken at the same time, and quality of life is assessed in all participants. At this point, depending on the participant's wishes, it is possible to perform sperm cryopreservation for fertility preservation before starting gender affirming hormonal treatment.
  Groups: tucking

SUMMARY:
Because gender-affirming hormone therapy (GAHT) can lead to fertility impairment, current guidelines and treatment recommendations require that patients be informed about the possibility of fertility preservation prior to initiating GAHT. A recent review by our working group analyzed the current data on fertility and fertility preservation in transgender and gender diverse people. Several studies were identified that evaluated semen quality before and during GAHT in trans women compared to reproductive men. All studies showed a significant reduction in semen quality even before GAHT. In addition, one study found evidence that constant wearing of tight underwear and tucking was associated with a reduction in motile sperm concentration to <5 mill/ml. Tucking is a method of avoiding crotch bulge through the penis and testicles by placing the penis backwards between the legs and optionally pushing the testicles into the groin canals. These positions are fixed with tight-fitting underwear or gaffs. Whether tucking or the wearing of tight underwear is the determining factor for impaired semen quality even before the start of GAHT and whether there is reversibility remains unclear and will be investigated in the present study.

The study is designed as a prospective case-control study with a total sample size of n = 40 trans women. All patients with gender incongruence presenting to the University Clinic for Gynecology, Endocrinology and Reproduction Innsbruck before starting GAHT are eligible to participate. Trans women (n = 20) who practice tucking or wear tight underwear will be included and trans women (n = 20) who do not practice tucking will be included as a control group. At Time 1, after 2-7 days of abstinence, all participants will provide a semen sample for a spermiogram, a venous blood sample will be taken, and quality of life will be assessed using a questionnaire. The frequency and duration of tucking or wearing tight underwear, ejaculation frequency, demographic data such as BMI, nicotine use, alcohol and drug use, medication use, underlying medical conditions, previous surgeries, etc. are also recorded.

Participants in the study group are then asked to abstain tucking for at least 73 days. After 2-7 days of sperm abstinence, another semen sample is taken at time 2, a venous blood sample is taken, and quality of life is assessed. At this point, depending on the participant's wishes, there is the option of sperm cryopreservation for fertility preservation prior to starting GAHT.

Spermiograms are performed under standardized conditions according to current WHO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Female transgender patients between the ages of 18 to 50 years of age who are seen at the University Clinic for Gyn. Endocrinology and Reproductive Medicine of the Medical University of Innsbruck. Patients must have met the eligibility and readiness criteria for gender-affirming hormone therapy

Exclusion Criteria:

* Ongoing GAHT gender affirming genital surgery Hypogonadism Diabetes mellitus Cystic Fibrosis Varicocele Cryptorchism Post-sterilization Incapacity to consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female gender identity
Study Population: Female transgender patients between the ages of 18 to 50 years of age who are seen at the University Clinic for Gyn. Endocrinology and Reproductive Medicine of the Medical University of Innsbruck. Patients must have met the eligibility and readiness criteria for gender-affirming hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
semen concentration | 3 months
  Semen quality defined by semen concentration, motility and total volume with and without tucking
semen motility | 3 months
  Semen quality defined by semen concentration, motility and total volume with and without tucking
semen total volume | 3 months
  Semen quality defined by semen concentration, motility and total volume with and without tucking

SECONDARY OUTCOMES:
LH | 3 months
  hormone levels with and without tucking
FSH | 3 months
  hormone levels with and without tucking
estradiol | 3 months
  hormone levels with and without tucking
testosterone | 3 months
  hormone levels with and without tucking
quality of life assessment | 3 months
  measured with the questionnaire "iTransQoL"

CONTACTS AND LOCATIONS:
Locations (1):
- University clinic for Gynecological Endocrinology and Reproductive Medicine Department of Gynecology Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided